CLINICAL TRIAL: NCT01971229
Title: Assessment of Insulin Response Following Ingestion of a Carbohydrate/Whey Protein Drink. A Cross-over Randomized Double Blind Study.
Brief Title: Gastric Emptying and Insulin Response to Test Drink
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Franco Carli (Other)
Responsible Party: Sponsor-Investigator, Franco Carli, Professor, Department of Anesthesia, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 13-168-BMA
Record Dates: First submitted 2013-10-23; First posted 2013-10-29 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Insulin Resistance
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Carbohydrate (Sham Comparator): Patients in this arm will drink a 425 mL 100% clear apple juice (carbohydrate 50 g, 700 mOsmol). 1.5 g of acetaminophen will be dissolved in the beverage for determination of gastric emptying.
  Interventions: Other: Carbohydrate based drink; Other: Whey protein based drink
- Whey Protein (Active Comparator): Patients in this arm will drink a 330 mL Boost fruit flavoured clear beverage (whey protein 12.2 g, carbohydrate 50 g, 700 mOsmol).1.5 g of acetaminophen will be dissolved in the beverage for determination of gastric emptying.
  Interventions: Other: Carbohydrate based drink; Other: Whey protein based drink

INTERVENTIONS:
Other: Carbohydrate based drink — After consumption of the test drink to record the insulin response and gastric emptying.
Other: Whey protein based drink — After consumption of the test drink to record the insulin response and gastric emptying.

SUMMARY:
Surgery is a stress on the body and recovering well after surgery is very important to patients and their doctors. It is therefore important to prepare patient's bodies for the stress of surgery, and one way to do this is to provide proper nutrition. In the past, patients were asked to prepare for surgery by fasting from midnight before surgery. Today, it is known that this practice is not beneficial to patient's recovery. In fact, it has been recognized that drinking a sugary beverage (e.g., juice) before surgery stimulates the production of insulin, which is a hormone that helps make the proteins needed for wound healing after surgery. This is currently practiced at the MUHC. It might also be beneficial, however, to drink a beverage that contains sugar and whey proteins (a protein isolated from milk) before surgery. In fact, whey proteins stimulate insulin and may also have the added benefit of improving muscular strength. In this study, investigators will measure the level of insulin produced after drinking a carbohydrate (i.e., sugar)-whey protein beverage to determine how it compares to the level of insulin produced after drinking the sugary beverage used at the MUHC.

DETAILED DESCRIPTION:
It is hypothesized that the increase in plasma insulin following a mixed carbohydrate whey protein drink is significantly greater than that elicited by a carbohydrate drink.

ELIGIBILITY:
Inclusion Criteria:

- Healthy volunteer

Exclusion Criteria:

* diabetes,
* neurological disorders
* chronic kidney failure
* chronic liver disease
* disorders of gastric motility
* gastro-esophageal reflux
* achalasia
* gastroparesis
* intestinal obstruction
* previous abdominal surgery
* lactose intolerance
* body mass index below 17 or above 29
* allergy to acetaminophen.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-12; Primary Completion 2014-10 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Insulin response to a test meal | Change over 3 hours
  Patients will consume a carbohydrate or a whey protein based drink and their insulin response will be monitored every 30 minutes for 3 hours.

SECONDARY OUTCOMES:
Gastric emptying | Change over 3 hours
  The acetaminophen absorption test, as an indirect assessment of gastric emptying.Since gastric emptying is the rate-limiting step in delivering the drug to its absorption site, it is believed that the rate of appearance of acetaminophen in the blood reflects the rate of gastric emptying.
  Blood samples will be collected every 30 minutes for 3 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Franco Carli, MD, Principal Investigator — Montreal General Hospital
Locations (1):
- Montreal General Hospital, Montreal, Quebec, Canada